CLINICAL TRIAL: NCT02169869
Title: Immediate Postplacental Intrauterine Device Insertion in High-risk Patient Populations
Brief Title: Immediate Postplacental IUD Insertion
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in local healthcare policies and practices
Sponsor: Oregon Health and Science University (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Principal Investigator, Jeffrey Jensen, Research Director, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: OHSU IRB #10473
Record Dates: First submitted 2014-06-19; First posted 2014-06-23 (Estimated); Results first posted 2019-05-01 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Contraception
Keywords: intrauterine device, postpartum, contraception, Mirena, Paragard, intrauterine system

STUDY DESIGN:
Intervention Model Description: randomized-controlled trial
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate postplacental IUD insertion (Experimental): Women randomized to the immediate postplacental IUD group will receive their IUD within 60 minutes of placental delivery.
  Interventions: Device: Mirena; Device: Paragard
- 6 weeks postpartum IUD insertion (Active Comparator): Subjects who are randomized for IUD insertion at their postpartum visit will be assisted in scheduling a postpartum visit and IUD placement with their usual obstetrical care provider.
  Interventions: Device: Mirena; Device: Paragard

INTERVENTIONS:
Device: Mirena — A radio-opaque T-shaped polyethylene device containing 52mg of levonorgestrel dispersed in polydimethylsiloxane on its stem. The progestin is released at a rate of 15 mcg per day.
  Other Names: levonorgestrel intrauterine system
Device: Paragard — A T-shaped polyethylene device with 380 mm2 of exposed surface area of fine copper wire wound around its arms and stem. Barium sulfate has been added to the polyethylene frame to make the device radio-opaque. A 3-mm plastic ball is located at the base of the IUD, through which the polyethylene monofilament string passes.
  Other Names: Copper T380A IUD

SUMMARY:
The study will be a randomized clinical trial. Women with less than 10 prenatal visits and/or 2 or more no show visits who desire an Intrauterine Device (IUD) will be considered for enrollment. If consented and meet inclusion criteria, they will be randomized after delivery to receive an IUD immediately postplacental or at their routine postpartum visit.

Women who plan to deliver a live birth singleton via vaginal or cesarean delivery at Oregon Health and Science University (OHSU) hospital will be considered for inclusion in the study. Women who desire an IUD for postpartum contraception will be approached for study participation. The postpartum contraception plan is routinely documented during their prenatal course. It is also addressed by the obstetrical team upon admission to Labor & Delivery at OHSU. The obstetrical team will identify subjects who present in labor who meet the criteria of poor prenatal clinic attendance and express interest in intrauterine contraception. Immediately after vaginal or cesarean delivery, consented subjects will be randomized to immediate postplacental IUD placement or IUD placement at their routine postpartum visit. Women randomized to the immediate postplacental IUD group will receive their IUD within 60 minutes of placental delivery. Prior to discharge from the hospital women who received a postplacental IUD will be assisted in scheduling a routine postpartum visit with their primary provider. Subjects who are randomized for IUD insertion at their postpartum visit will be assisted in scheduling a postpartum visit and IUD placement with their usual obstetrical care provider. All subjects in the delayed group will be provided with contact information for the Women's Health Research Unit (WHRU) at OHSU. If a subject cannot obtain an IUD at her usual place of care, the device will be placed at no cost through the WHRU.

At 3 months after delivery, all subjects will be contacted by phone, text, or email to complete a questionnaire to determine whether they have had a known expulsion, pregnancy, or elective IUD removal. The questionnaire will include questions regarding ease of placement and overall satisfaction with the timing of placement. Subjects will be compensated for their participation in the study after the 3 month contact.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18 yo or older
* Singleton pregnancy at ≥32 weeks gestation at time of enrollment
* Voluntarily requesting either copper T380A or levonorgestrel IUD (LNG-IUS) placement for postpartum contraception
* English or Spanish speaking
* Able to give consent and agree to the terms of the study
* Less than 10 prenatal visits or 2 or more no show visits
* Since IUDs are not on our hospital formulary, the patient must qualify for a Long Acting Reversible Contraceptive (LARC) IUD (this includes all Oregon Health Plan (OHP) or Citizen/Alien Waived Emergent Medical (CAWEM) insured patients or women with income <300% of the federal poverty line).

Exclusion Criteria:

* Anatomic uterine abnormalities that prevent proper fundal placement of IUD (obstructive myomata, bicornuate, septate, etc)
* Chorioamnionitis (also consider other risk factors such as prolonged rupture of membranes >18 hours, prolonged labor >24 hours, fever >38C)
* Puerperal sepsis
* Unresolved postpartum hemorrhage
* Extensive genital trauma
* Current incarceration
* Known or suspected untreated endocervical gonorrhea, chlamydia
* Wilson's disease, copper allergy (Paragard only)
* Known or suspected cervical or endometrial cancer or pelvic tuberculosis
* Current breast cancer (LNG-IUS only)
* Systemic lupus erythematosus (SLE) with severe thrombocytopenia (Paragard only)
* Trophoblastic disease (benign or malignant)
* AIDS not stable on antiretroviral

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2014-09; Primary Completion 2017-01-31 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Jensen, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Immediate Postplacental IUD Insertion | 6 Weeks Postpartum IUD Insertion
Started | 17 | 16
Completed | 17 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Postplacental IUD Insertion | 6 Weeks Postpartum IUD Insertion | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 16 | 33
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 16 | 33
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 17 | 16 | 33

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With an IUD at 3 Months Postpartum
Description: Subjects were contacted at 3 months after delivery. Comparison of the proportion of women randomized to placement of IUD within 60 minutes of placental delivery or at their 6-week routine postpartum visit who report having an IUD in place at 3 months after delivery.
Time Frame: 3 months postpartum (after delivery)
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Postplacental IUD Insertion | 6 Weeks Postpartum IUD Insertion
Number analyzed (Participants) | 17 | 16
Participants | 12 | 5

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Immediate Postplacental IUD Insertion | 6 Weeks Postpartum IUD Insertion
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 0/17 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-16): https://cdn.clinicaltrials.gov/large-docs/69/NCT02169869/Prot_SAP_000.pdf